CLINICAL TRIAL: NCT02886624
Title: Short Duration Therapy of Acute Hepatitis C Genotypes 1 or 4: Efficacy and Tolerability of Grazoprevir 100mg/Elbasvir 50mg During 8 Weeks
Brief Title: Short Duration Therapy of Acute Hepatitis C Genotypes 1 or 4
Acronym: SAHIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 50
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Acute Hepatitis C; HIV
MeSH Terms: interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Grazoprevir/Elbasvir (Experimental): Once-daily, oral grazoprevir/elbasvir combination therapy at fixed-dose (100mg/50mg) for 8 weeks
  Interventions: Drug: Grazoprevir/Elbasvir

INTERVENTIONS:
Drug: Grazoprevir/Elbasvir — Once-daily, oral grazoprevir/elbasvir combination therapy at fixed-dose (100mg/50mg) for 8 weeks
  Other Names: Zepatier

SUMMARY:
The purpose of this study is to assess the rate of sustained virological response (SVR) 12 weeks after 8-week oral treatment with grazoprevir 100mg/elbasvir 50mg (MRK-combo) in patients with acute hepatitis C genotype1 or 4.

DETAILED DESCRIPTION:
Increasing rates of acquisition of HCV in men who have sex with men (MSM) have been reported since 2001 in Western European countries and particularly in France. Observational studies have recently reported that HIV-infected gay and bisexual men with sexually transmitted hepatitis C have shown unexpectedly rapid liver disease progression in a relatively short period of time.

It is therefore admitted that, in the absence of a spontaneous HCV clearance within 3 months of acute HCV infection, treatment should be initiated. Pegylated interferon in combination with weight-adapted ribavirin is still recommended as the treatment of choice for all HCV genotypes in an acute setting. For patients developing a rapid virologic response, treatment duration of 24 weeks is recommended. If antiviral therapy was initiated within 24 weeks after diagnosis, sustained virologic response rates of 60 to 80% have been observed at the price of a high side effects burden.

However, short course therapies with new direct acting antivirals are likely to be safer and more efficient. But their efficacy in acute hepatitis C has still to be established. To date, US- and Europe- based trials are ongoing in this setting with the association of sofosbuvir and ribavirine, sofosbuvir / ledipasvir or sofosbuvir / simeprevir, for a duration of 4, 6, 8 or 12 weeks. Preliminary results are very diverse, with SVR12 ranging from 56% to 95%. MSD has been evaluating the efficacy and safety of a double drug combination (grazoprevir + elbasvir) in HIV-infected patients which exhibits paramount efficacy and excellent tolerance in a diverse range of genotypes, including 1 and 4 HCV strains, which are those mainly encountered in the French acute HCV epidemics in MSM. This association has the potential to be used for short treatment duration especially with regards to the fact that patients will have no fibrosis at the time of treatment initiation. This MRK-combo would therefore be an ideal candidate for treating acute hep C due to GT1 or 4 in a "test and treat" approach in high-risk population such as MSM.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years.
2. A recent acute HCV infection [defined by (i) detectable HCV RNA within 6 months after a negative HCV RNA or HCV serology test OR (ii) detectable HCV RNA and acute clinical hepatitis within 5 months prior to screening visit (ALT ≥250 IU/L with normal ALT within the preceding 8 months OR ALT ≥500 IU/L with either no measured ALT or with abnormal ALT within the preceding 8 months)] or reinfection [defined by documented de novo infection after prior clearance post-treatment (defined by one negative HCV RNA ≥6 months after end of treatment) or spontaneously (defined by two negative HCV RNA a minimum of 6 months apart OR documented infection with a new viral strain, confirmed by phylogenetic or genotypic analysis)] within 5 months prior screening OR (iii) patients having reported a risk factor for HCV contamination (traumatic sexual intercourse, intranasal, rectal or intravenous drug use) ≥6 months AND presenting a negative HCV RNA or HCV serology test within 12 months.
3. Infection with HCV genotype 1 or 4 (confirmed at screening visit or by using a previous biological test performed 1 to 4 weeks before week 0).
4. Plasma HCV-RNA ≥ 1000 IU/mL (confirmed at screening visit or by using a previous biological test performed 1 to 4 weeks before week 0).
5. Confirmed HIV infection (only for HIV co-infected patients).
6. Without HIV treatment or with an authorized stable HIV treatment for at least two weeks (only for HIV co-infected patients).
7. Body weight ≥40 kg and ≤125 kg.
8. Female patients with child-bearing potential and their heterosexual partners must use adequate contraception from the date of screening until 30 days after administration of the last dose of study drug. Male participants must agree to consistently and correctly use a condom, while their female partner must use adequate contraception from the date of screening until 30 days after administration of the last dose of study drug.
9. Informed and signed consent.
10. Patients with Health insurance (Sécurité Sociale or Couverture Médicale Universelle).

Exclusion Criteria:

1. Opportunistic infections (stage C), active or occurred within 6 months prior to baseline.
2. Primary HIV infection.
3. Co-infection with Hepatitis B virus (HBsAg-positive) without appropriate treatment (TDF or TAF) for at least 2 weeks.
4. Confirmed cirrhosis (before acute HCV diagnosis).
5. Any other causes of acute hepatitis.
6. Pregnant or breast-feeding women.
7. Liver transplant recipients.
8. Evolutive malignancy.
9. Patients with a history of non-adherence, who will be at risk of being unable to respect the study follow-up timetable.
10. Patients participating in another clinical trial (with an experimental treatment) or within an exclusion period of a previous clinical trial at screening.
11. Patients under legal gardianship or incarcerated.
12. Hemaglobulin <10 g/dL (female) or <11g/dL (male).
13. Platelet count <50,000/mm3.
14. Neutrophil count < 750/mm3.
15. Other antiretroviral drugs than those allowed in the study.
16. Contra-indications to grazoprevir and/or elbasvir or to any of the excipients listed in the summary of the product characteristics.
17. Contra-indicated treatment likely to interfere with the study drugs as listed in the summary of the product characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karine Lacombe, MD, PhD, Principal Investigator — Hôpital Saint-Antoine, Service des maladies infectieuses et tropicales
Locations (6):
- France (6):
  - CHU de Lyon, Lyon
  - CHU de Nice, Nice
  - Hôpital Saint-Antoine, Paris
  - Hôpital La Pitié-Salpêtrière, Paris
  - Hôpital Bichat, Paris
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: Yes
All data are available as IPD. An official request must be made to the Principal Investigator. The request will be reviewed by the Scientific Committee. If approved, data will be exchanged according to European Union General Data Protection Regulation.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data are available as of January 1, 2020 and will be available for request until December 31, 2025.
Access Criteria: Please contact the Principal Investigator for further details.

REFERENCES:
- [Background] Gambotti L, Batisse D, Colin-de-Verdiere N, Delaroque-Astagneau E, Desenclos JC, Dominguez S, Dupont C, Duval X, Gervais A, Ghosn J, Larsen C, Pol S, Serpaggi J, Simon A, Valantin MA, Velter A; Acute hepatitis C collaborating group. Acute hepatitis C infection in HIV positive men who have sex with men in Paris, France, 2001-2004. Euro Surveill. 2005 May;10(5):115-7. PMID 16077209
- [Background] Fierer DS, Dieterich DT, Fiel MI, Branch AD, Marks KM, Fusco DN, Hsu R, Smith DM, Fierer J. Rapid progression to decompensated cirrhosis, liver transplant, and death in HIV-infected men after primary hepatitis C virus infection. Clin Infect Dis. 2013 Apr;56(7):1038-43. doi: 10.1093/cid/cis1206. Epub 2012 Dec 21. PMID 23264364
- [Background] European AIDS Treatment Network (NEAT) Acute Hepatitis C Infection Consensus Panel. Acute hepatitis C in HIV-infected individuals: recommendations from the European AIDS Treatment Network (NEAT) consensus conference. AIDS. 2011 Feb 20;25(4):399-409. doi: 10.1097/QAD.0b013e328343443b. No abstract available. PMID 21139491
- [Background] Rockstroh JK, Nelson M, Katlama C, Lalezari J, Mallolas J, Bloch M, Matthews GV, Saag MS, Zamor PJ, Orkin C, Gress J, Klopfer S, Shaughnessy M, Wahl J, Nguyen BY, Barr E, Platt HL, Robertson MN, Sulkowski M. Efficacy and safety of grazoprevir (MK-5172) and elbasvir (MK-8742) in patients with hepatitis C virus and HIV co-infection (C-EDGE CO-INFECTION): a non-randomised, open-label trial. Lancet HIV. 2015 Aug;2(8):e319-27. doi: 10.1016/S2352-3018(15)00114-9. Epub 2015 Jul 9. PMID 26423374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between May 31, 2017 and August 20, 2019. Recruitment took place at 6 university hospitals in France (Paris, Lyon, and Nice). 33 individuals were assessed for eligibility and 3 did not meet inclusion criteria.
Period: 8-week Treatment
Arm/Group | Grazoprevir/Elbasvir
Started | 30
Completed | 30
Not Completed | 0
Period: 12-week Post Treatment Follow-up
Arm/Group | Grazoprevir/Elbasvir
Started | 30
Completed | 29
Not Completed | 1
Not completed — Death | 1
Period: 48-week Post Treatment Follow-up
Arm/Group | Grazoprevir/Elbasvir
Started | 29
Completed | 28
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [34 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 30
Co-infection with HIV [Count of Participants; unit: Participants] | 28

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Undetectable plasma HCV RNA (<12 IU/mL) 12 weeks post-treatment.
Time Frame: 12 weeks
Population: Intent-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 30
Participants | 28

2. Secondary Outcome: Virological Failure
Description: Number of patients harboring HCV (NS5A and NS3/4) resistance mutations 12 weeks post treatment
Time Frame: 12 weeks
Population: Intent-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 30
Participants | 1

3. Secondary Outcome: Treatment Adherence
Description: Number of patients missing study drug within the last four days during treatment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 30
Participants | 2

4. Secondary Outcome: Number of Participants With Undetectable HIV RNA
Description: Number of participants with undetectable HIV RNA at 12 weeks post treatment (in HIV-positive co-infected patients)
Time Frame: 12 weeks
Population: Out of 28 HIV-positive individuals, 27 had available data. All 27 participants analyzed had undetectable HIV RNA.
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 27
Participants | 27

5. Secondary Outcome: CD4 Cell Count
Description: CD4+ T cell count at 12 weeks post treatment (in HIV-positive co-infected patients)
Time Frame: 12 weeks
Population: Out of 28 HIV-positive individuals, 27 had available data.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 27
cells/mm^3 | 655 [488 to 829]

6. Secondary Outcome: Incidence of HCV Re-infection
Description: Number of patients with positive HCV RNA 48-weeks post treatment.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 28
Participants
  With phylogentically different strain | 2
  With phylogentically similar strain | 1

ADVERSE EVENTS:
Time Frame: Through evaluation of the primary endpoint (i.e. sustained virological response 12 weeks post treatment), an average of 20 weeks
Description: Patient reported (relayed by the treating physician) and laboratory adverse events (grading based in ANRS definitions) were provided. Deaths due to any cause were also provided.
Arm/Group | Grazoprevir/Elbasvir
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir/Elbasvir (N=30)
Suicide (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir/Elbasvir (N=30)
Syphilis (Infections and infestations) | 3 (3)
Primary HIV infection (Infections and infestations) | 1 (1)
Depressive disorder (Psychiatric disorders) | 1 (1)
Insomnia (General disorders) | 2 (2)
Secondary tremor from pulmonary heart disease (Cardiac disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other disorders of the nasal cavity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Xerostomia (Skin and subcutaneous tissue disorders) | 1 (1)
Dental caries (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth ache (Musculoskeletal and connective tissue disorders) | 1 (1)
Vesicular dermatitis of hands and feet (Skin and subcutaneous tissue disorders) | 1 (1)
Eczematous dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Chronic paronychia (Skin and subcutaneous tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Male erectile dysfunction (Reproductive system and breast disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Binge eating (Metabolism and nutrition disorders) | 1 (1)
Dysgeusia (Metabolism and nutrition disorders) | 1 (1)
Cramp or spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain localised to abdomen (Musculoskeletal and connective tissue disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Pain in knee joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Fatigue (General disorders) | 5 (6)
Insect bite (Injury, poisoning and procedural complications) | 1 (1)
Voluntary drug intoxication (Injury, poisoning and procedural complications) | 1 (1)
Mycoplasma genitalium (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02886624/Prot_SAP_000.pdf